CLINICAL TRIAL: NCT04398524
Title: A Phase II Study of Cemiplimab, an Anti-PD-1 Monoclonal Antibody, and ISA101b Vaccine in Patients With Recurrent/Metastatic HPV16 Positive Oropharyngeal Cancer Who Have Experienced Disease Progression With Prior Anti-PD-1 Therapy
Brief Title: A Phase II Study of Cemiplimab and ISA101b in Patients With Recurrent/Metastatic HPV16 Positive OPC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ISA Pharmaceuticals (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISA101b-OPC-03-19
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Squamous Cell Carcinoma of the Oropharynx
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): ISA101b 4 times plus cemiplimab every 3 weeks for up to 24 months
  Interventions: Drug: ISA101b

INTERVENTIONS:
Drug: ISA101b — ISA101b 4 times plus cemiplimab every 3 weeks for up to 24 months
  Other Names: Cemiplimab

SUMMARY:
This will be an open-label, phase 2 study in which subjects will receive ISA101b and cemiplimab.

DETAILED DESCRIPTION:
This study will assess the ability of ISA101b plus cemiplimab to improve Overall Response Rate in subjects who have progressed on prior anti-PD-1 therapy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age.
* Provide informed consent signed by study patient.
* Willing and able to comply with site visits and study-related procedures and requirements.
* Histologically confirmed recurrent or metastatic HPV16 positive OPC. Patients with squamous cell carcinoma of occult primary site, presenting with lymph node(s) limited only to the neck, are also eligible. Patients should have HPV16 positivity confirmed before being considered a candidate for this study.
* HPV16 genotyping as determined by a specified central reference laboratory. If local specific HPV16 genotype assessment has been performed, the patient can be enrolled if the result shows HPV16 positivity. Confirmation of HPV16 positive status will then subsequently have to be performed by the central laboratory.
* Patients who have received a minimum total dose of 600 mg of pembrolizumab or 960 mg of nivolumab or equivalent anti-PD-1 antibody with or without chemotherapy for only 1st or 2nd line recurrent/ metastatic HPV16 positive OPC. The last dose of anti-PD-1 must have been no more than 6 months prior to the first dose of study drug. Progressive disease (PD) must have been diagnosed during or after anti-PD-1 therapy (but not longer than 6 months after the last dose), and anti PD-1 therapy (as 1st or 2nd line for recurrent/metastatic HPV16 positive OPC) should have been the last treatment regimen that the patient received before entry into the current trial.
* At least one measurable lesion by CT or MRI per RECIST version 1.1 criteria. Target lesions may be located in a previously irradiated field if there is documented disease progression in that site.
* Eastern Cooperative Oncology Group performance status of 0 or 1.

Exclusion Criteria:

* Invasive surgery (defined as surgical intervention requiring general or spinal anesthesia and hospital admission) within 4 weeks prior to start of study treatment.
* Patients who, after progressing on anti-PD-1, received additional anti-cancer therapy (chemotherapy, radiotherapy, experimental TKI's, immunotherapy, anti-EGFR antibodies, surgery). The following palliative treatments are allowed:
* palliative radiotherapy (but NOT for target lesions)
* palliative surgery
* bone resorptive therapy such as bisphosphonates and denosumab but only if patients have been on stable doses for > 4 weeks prior to first dose of test treatment
* Patients who have permanently discontinued anti-cancer immune modulating therapies due to drug-related toxicity.
* Ongoing or recent (within 5 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments. The following are not exclusionary: vitiligo, childhood asthma that has resolved, endocrinopathies (such as hypothyroidism or type 1 diabetes) that require only hormone replacement, or psoriasis that does not require systemic treatment.
* Untreated or active primary brain tumor, central nervous system (CNS) metastases, leptomeningeal disease or spinal cord compression.
* Encephalitis, meningitis, organic brain disease (e.g. Parkinson's disease) or uncontrolled seizures in the year prior to first dose of study therapy.
* Known history of, or any evidence of interstitial lung disease, or active, non-infectious pneumonitis (in the past 5 years). A history of radiation pneumonitis in the radiation field is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate based on radiographic response | 20-25 monhts
  Measured by RECIST version 1.1.

CONTACTS AND LOCATIONS:
Locations (41):
- United States (8):
  - City of Hope National Medical Center, Duarte, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Anschutz Cancer Pavilion, Aurora, Colorado
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Providence Portland Medical Center, Portland, Oregon
- Belgium (3):
  - University Hospital Antwerp, Antwerp
  - University Hospital Ghent, Ghent
  - Centre Hospitalier Universitaire de Liege, Liège
- Czechia (3):
  - Clinic of Oncology, Olomouc
  - Institute of Radiation Oncology, Prague
  - University Hospital Motol, Clinic of Oncology, Prague
- France (7):
  - Saint Andre Hospital, Department of Oncology, Bordeaux
  - Leon Berard Center, Department of Medical Oncology, Lyon
  - CHU La Timone - La Timone Children's Hospital, Marseille
  - Georges Pompidou European Hospital, Paris
  - Jean Godinot Institute, Cancer Research Center, Reims
  - Paul Strauss Center, Strasbourg
  - Gustave Roussy Institute, Villejuif
- Germany (5):
  - University Hospital Cologne, Department of Otorhinolaryngology (ENT), Cologne
  - University Hospital Giessen and Marburg GmbH, Giessen
  - University Hospital Mannheim, Mannheim
  - Caritas Klinikum, Saarbrücken
  - University Hospital Ulm, Ulm
- Israel (2):
  - Hadassah Medical Center, Jerusalem
  - The Tel Aviv Sourasky Medical Cente, Tel Aviv
- Italy (5):
  - Università degli Studi di Brescia, Brescia
  - European Institute of Oncology (IEO), IRCCS, Department of Otolaryngology and Facial Cervix Surgery, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - National Cancer Institute - IRCCS, Naples
  - Institute of Cancer Research and Treatment of Candiolo, Turin
- Spain (5):
  - Hospital Clinic of Barcelona, Barcelona
  - University Hospital Vall d'Hebron, Barcelona
  - Catalan Institute of Oncology, Hospital Duran i Reynals, Department of Oncology, L'Hospitalet de Llobregat
  - University Clinic of Navarra - Madrid, Madrid
  - University Clinic of Navarra, Pamplona
- United Kingdom (3):
  - Guy's Hospital, London
  - Royal Marsden Hospital, London
  - Royal Marsden Hospital - Sutton, Sutton